CLINICAL TRIAL: NCT02670707
Title: Randomization of Cytarabine Monotherapy Versus Standard-of-Care Vinblastine/Prednisone for Frontline Treatment of Langerhans Cell Histiocytosis (TXCH LCH0115)
Brief Title: Vinblastine/Prednisone Versus Single Therapy With Cytarabine for Langerhans Cell Histiocytosis (LCH)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Olive Eckstein, Assistant Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-37718 TXCH LCH0115
Record Dates: First submitted 2016-01-04; First posted 2016-02-02 (Estimated); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Langerhans Cell Histiocytosis
Keywords: vinblastine; prednisone; cytarabine; Langerhans Cell Histiocytosis (LCH)
MeSH Terms: conditions — Histiocytosis, Langerhans-Cell | interventions — Cytarabine; Vinblastine; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cytarabine ("experimental") arm (Experimental): On this arm, patients will receive single therapy with cytarabine.
  Interventions: Drug: Cytarabine
- Vinblastine/prednisone ("standard") arm (Active Comparator): On this arm, patients will receive standard-of-care therapy with vinblastine and prednisone.
  Interventions: Drug: Vinblastine/prednisone

INTERVENTIONS:
Drug: Cytarabine — Cytarabine 100 mg/m^2/day IV for five consecutive days. This five-day cycle will be repeated every 21 days for a total of four cycles for all patients regardless of response. Each new cycle may not begin until absolute neutrophil count (ANC) is ≥ 750/mcL and platelet count is ≥ 75,000/mcL.
  Other Names: cytosine arabinoside (ara-C)
  Arms: Cytarabine ("experimental") arm
Drug: Vinblastine/prednisone — Vinblastine/Prednisone +/- 6-mercaptopurine based on risk category. Patients with high-risk organ involvement (liver, spleen, hematopoeitic system) will receive 6-mercaptopurine during Continuation Therapy as this is the current standard of care treatment.
  Vinblastine 6 mg/m^2/dose IV push weekly for patients ≥ 12 months of age. Vinblastine will be dosed at 3 mg/m^2/dose for patients under 6 months of age, and dosed at 4.5 mg/m^2/dose for patients 6 months of age to 11.99 months of age.
  Prednisone (or prednisolone) 20 mg/m2/dose by mouth twice a day
  Other Names: Velban/Deltasone
  Arms: Vinblastine/prednisone ("standard") arm

SUMMARY:
Langerhans Cell Histiocytosis (LCH) is a type of cancer that can damage tissue or cause lesions to form in one or more places in the body. Langerhans cell histiocytosis (LCH) is a cancer that begins in LCH cells (a type of dendritic cell which fights infection). Sometimes there are mutations (changes) in LCH cells as they form. These include mutations of the BRAF gene. These changes may make the LCH cells grow and multiply quickly. This causes LCH cells to build up in certain parts of the body, where they can damage tissue or form lesions.

For most patients with LCH, standard-of-care vinblastine/prednisone are used as front-line therapy while cytarabine therapy has been used as therapy for patients who develop recurrence. No alternate treatment strategy has been developed for frontline therapy in LCH.

The purpose of this research study is to compare previously used vinblastine/prednisone to single therapy with cytarabine for LCH. We will evaluate the utility of an imaging study called a positron emission tomography (PET) scan to more accurately assess areas of LCH involvement not otherwise seen in other imaging studies as well as response to therapy. We also want to identify if genetic and other biomarkers (special proteins in patient's blood and in patient's cancer) relate to the response of patients LCH to study treatment.

DETAILED DESCRIPTION:
To be eligible to participate in this study, patients physician must have determined that they have LCH which is not treatable by surgical intervention or observation alone. If patient chooses to participate in this study, they will be assigned randomly (like flipping a coin) to one of two LCH chemotherapy treatment groups. A computer will randomly determine if they will begin to receive vinblastine/prednisone treatment or cytarabine treatment. Patient will have an equal chance (50%) to receive vinblastine/prednisone or to receive cytarabine. Neither the patient nor their doctor will be able to choose the group assignment, but the patient and their study doctor will know which treatment they are receiving.

The patient will need to have the following tests, exams, or procedures. Most of these are part of regular cancer care and may be done even if the patient does not want to join this study. Some of them may not need to be repeated if they have had them done recently. The patient's doctor will tell them which ones they need to repeat.

* History and Physical
* Blood tests
* Urine tests
* Biopsy to confirm diagnosis
* Bone Marrow biopsy/aspirate (if patient is less than 2 years old or for any patient clinical concern for bone marrow disease)*
* Lumbar puncture for spinal fluid tests (if patient has disease in pituitary gland or brain)

  * The bone marrow sample procedure is as follows: The skin above the hipbone will be made numb. This area will then be sterilized and a small incision will be made. A bone marrow needle will be inserted into the hipbone and bone marrow will be withdrawn. Patient will sign a separate consent that explains this procedure in more detail.

We will also do x-rays and scans of the inside of the body. These scans may include chest and bone x-rays, ultrasound, computerized tomography (CT), magnetic resonance imaging (MRI) and/or positron emission tomography (PET). The specific tests depend on age, sites of LCH and other clinical factors. An ultrasound is a sound wave machine that uses a computer to make pictures of the tissues of the body. A CT is an x-ray machine that uses a computer to make pictures of the organs of the body. An MRI is a scan which uses a magnetic machine to make pictures of the inside of the body. A PET scan is an x-ray technique that uses a sugar solution that you drink to see activity inside the body. The PET and CT scans will look at where the LCH is in the body.

If tests show that the patient can participate in this study and they choose to participate, treatment will begin based on randomization to either the cytarabine ("experimental") arm or the vinblastine/prednisone ("standard") arm as described below.

Patient will have a history and physical and blood tests before each cycle. The cancer drugs will be given to the patient intravenously (IV). An IV is a tube placed inside a vein to give medicine to the patient. If at anytime during the study the cancer gets worse, the patient will be taken off the study treatment.

1. Cytarabine ("experimental") arm

   Initial therapy I (Weeks 1-6)

   • Cytarabine for five consecutive days. This five-day cycle will be repeated every 21 days for a total of two cycles.

   Patient will have scans to see how the LCH responded to the treatment during week 6. Patients who have Complete Response (CR), Partial Response (PR), or Stable Disease (SD) at the end of Initial Therapy I, will proceed to Initial Therapy II (Weeks 7-12). Patients who have PR or SD at the end of Initial Therapy I will require reassessment again at the end of Initial Therapy II. Patients who have CR at the end of Initial Therapy I do not require disease reassessment again until Continuation Week 24.

   Initial therapy II (Weeks 7-12)

   • Cytarabine for five consecutive days. This five-day cycle will be repeated every 21 days for a total of two cycles.

   Patient will have scans to see how the LCH responded to the treatment during week 12 (unless they had no active disease at week 6). If the patient had LCH in their bone marrow (BM) at the beginning of the study, they will have another BM biopsy. If the cancer is stable and does not respond to therapy by Week 12, the patient will be taken off the study treatment. If the patient has no evidence of active disease at this time they will proceed to Continuation therapy.

   Continuation therapy (Weeks 13-52)

   • Cytarabine for five consecutive days. This five-day cycle will be repeated every 28 days for 10 additional cycles to complete one year of therapy

   Patient will have scans to see how the LCH responded to the treatment at Week 24 and at the end of therapy. If the patient had LCH in their bone marrow (BM) at the beginning of the study, they will have another BM biopsy.
2. Vinblastine/prednisone ("standard") arm

Initial therapy I (Weeks 1-6)

* Prednisone given by mouth two times a day daily on days 1-28 AND
* Vinblastine will be given IV (into a vein) one day a week for 6 weeks

Patient will have scans to see how the LCH responded to the treatment after week 6. If the patient had LCH in their bone marrow (BM) at the beginning of the study, they will have another BM biopsy. If the disease is completely gone by Week 6, patient will proceed to Continuation therapy. If the disease is only partly gone or unchanged patient will receive additional therapy with Initial therapy II.

Patient will have scans to see how the LCH responded to the treatment during Week 12 and if they had LCH in their bone marrow (BM) at the beginning of the study, they will have another BM biopsy.

Initial therapy II (Weeks 7-12, given only if the patient does not have evidence of active disease by Week 6)

* Prednisone by mouth on the first three days of each week during weeks 7-12 AND
* Vinblastine IV weekly during weeks 7-12

If the disease is gone or better after this additional therapy Continuation therapy will begin.

Continuation therapy

* Prednisone by mouth twice daily day on days 1-5 every 3 weeks AND
* Vinblastine IV once every 3 weeks
* 6-Mercaptopurine by mouth daily NOTE: Only high risk patients will receive 6-Mercaptopurine

Patient will have scans to see how the LCH responded to the treatment at Week 24 and at the end of therapy. If the patient had LCH in their bone marrow (BM) at the beginning of the study, they will have another BM biopsy.

STUDY FOLLOW-UP: Patient will be in this study for 5 years after completion of their therapy. The doctors will exam the patient at 1 month, 3 months, 6 months, 9 months, 12 months, then at 18 and 24 months, then yearly until 5 years after the patient is taken off treatment. At these visits the patient may have routine blood tests, scans, and the biology tests.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must have biopsy-confirmed diagnosis of Langerhans cell histiocytosis.
2. Patient must be between 0-21 years of age.
3. Patient must have a Karnofsky performance score ≥ 50% or Lansky performance score ≥ 50%.

Exclusion Criteria:

1. Patient may not have received any prior systemic cytotoxic or other chemotherapies for LCH or any other malignant disorder prior to the initiation of protocol therapy on TXCH LCH0115 with the exception of:

   Steroid pretreatment: Systemic glucocorticosteroids (prednisone, methylprednisone, dexamethasone, etc.) for less than or equal to 120 hours (5 days) in the 7 days prior to initiating protocol therapy or for less than or equal to 336 hours (14 days) in the 28 days before the initiation of protocol therapy does not affect eligibility. The dose of steroid previously given does not affect eligibility. Patients who have only received surgical or radiation therapy, intralesional injection of steroids, inhalational steroids, systemic mineralocorticoids (hydrocortisone), or topical steroids may also be enrolled.
2. Patient may not have disease limited to a single skin or bone site, with the following exceptions:

   * Central Nervous System (CNS) risk lesions/special site disease: patients with single bone sites that are CNS-risk (sphenoid, mastoid, orbital, zygomatic, ethmoid, maxillary, or temporal bones, the cranial fossa, pituitary gland or neurodegenerative disease) or are "special sites" (odontoid peg, vertebral lesion with intraspinal soft tissue extension) require systemic therapy as standard of care and thus are eligible for the study.
   * Functionally critical lesions: A single lesion not described above which may cause "functionally critical anatomic abnormality" wherein attempts at local therapy (such as surgical curettage or radiation) would cause unacceptable morbidity. These patients may be enrolled with written approval of the Coordinating Center PI or Vice-Chair and documentation of the rationale justifying systemic therapy.
   * Asynchronous multisite LCH presentation: A patient may also have any single site of disease involvement at the time of enrollment if they previously had at least one other site of LCH disease in the past (which may have been treated with local therapy/surgery as described), as long as no systemic therapy was previously given per protocol guidelines.
3. Patient may not have severe renal disease (creatinine greater than 3 times normal for age OR creatinine clearance < 50 ml/m2/1.73m^2).
4. Patient may not have severe hepatic disease (direct bilirubin greater than 3 mg/dl OR aspartate aminotransferase (AST) greater than 500 IU/L), unless hepatic injury is due to LCH.
5. Female patients may not be pregnant or breastfeeding.
6. Patients of reproductive potential not willing to use an adequate method of birth control for the duration of the study.
7. Patients who are HIV positive may not be enrolled.

NOTE: Patients excluded for laboratory abnormalities or performance score only may be enrolled on the study with written approval from the Coordinating Center PI or Vice-Chair.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 124 (Estimated)
Dates: Start 2016-03-07 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Time to determine 1-year event-free survival (EFS) of patients treated with cytarabine monotherapy for LCH, compared directly with that of standard-of-care vinblastine/prednisone (Events include progression of LCH, relapse, or death). | up to 60 months
  A Kaplan-Meier curve will be used to compare event-free survival between treatment groups. Curves will be compared using the log-rank statistic. Patients will be followed for up to 5 years after one year of therapy. Patients who have not had the event by the 5-year mark will be censored observations. Patients who are lost to follow-up without having an event will be censored at the time of last contact. Statistical significance will be assessed at the 0.05 level.
  A Cox proportional hazards model will also be used to estimate the Hazards Rate for combined events in the Cytarabine group versus standard therapy. A multiple regression model will also be used to estimate the adjusted HRs for genotype and baseline risk of death (high vs. low).

SECONDARY OUTCOMES:
Durable responses with 2-year and 5-year EFS and OS of the patients treated with cytarabine versus vinblastine/prednisone for LCH. | 2-years and 5-years post treatment
  Overall disease response at each timepoint will be assigned based on the lesion or organ system with worst response. For disease response not defined by the criteria included in the protocol, guidelines established in the RECIST criteria will be used.
Number of toxicities (including psychosis, hypertension, neuropathy, fever, headache) in the patients treated with cytarabine versus vinblastine/prednisone for LCH. | up to 60 months after completion of therapy
  Toxicity will be graded by the NCI Common Toxicity Criteria Version 5.0.
Rate at which patients achieve non-active disease on cytarabine versus vinblastine/prednisone therapy. | up to 60 months after completion of therapy
  RECIST criteria will be used for assessing disease response
Time to eradication of BRAF-V600E cells or other LCH-defining mutation | within 6-24 weeks of therapy initiation
  This will be quantified by quantitative real-time PCR.
Number of patients who have 18-FDG PET/CT positivity in identifying high-risk organ (liver, spleen, or bone marrow) involvement and correlation of PET/CT response with presence of disease activity as well as presence of circulating cells with BRAF-V600E. | up to 60 months after completion of therapy
  For disease response not defined by the criteria included in the protocol, guidelines established in the RECIST criteria will be used.
RECIST criteria and terminology in conjunction with metabolic PET imaging (where applicable) to assess disease response to therapy. | up to 60 months after completion of therapy
  This trial will utilize RECIST criteria for assessing disease response, which uses standard oncology response criteria terminology. Using RECIST terminology, we define response criteria for organs that may not have measurable lesions (i.e. bone marrow) but are clearly critical sites of disease. In addition, definitions of response in terms of metabolic activity from PET scans will also be prospectively analyzed based on prior retrospective radiologic reviews.
Number of risk factors for and time to development of diabetes insipidus and neurodegenerative disease. | up to 60 months after completion of therapy
  Evaluation of CNS+ site involvement at start of therapy, somatic BRAFV600E mutation status and measurable peripheral/marrow levels, ethnicity, age at onset, and extent of disease in predicting risk of neurodegenerative disease and/or pituitary involvement.
Storage of serial samples | up to 60 months after completion of therapy
  To store serial samples (viable WBCs, plasma, tumor, bone marrow, cerebrospinal fluid) for future correlative biology studies.

CONTACTS AND LOCATIONS:
Overall Officials: Olive Eckstein, MD, Study Chair — Baylor College of Medicine
Locations (11):
- United States (11):
  - Stanford Children's Hospital, Lucile Packard Children's Hospital, Palo Alto, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Nationwide Children's Hospital, Columbus, Ohio
  - Lehigh Valley Health Network- Cedar Crest, Allentown, Pennsylvania
  - Dell Children's Medical Center, Austin, Texas
  - Cook Children's Health Care System, Fort Worth, Texas
  - Texas Children's Hospital, Houston, Texas
  - Vannie Cook Children's Clinic, McAllen, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas
  - Children's Hospital of The King's Daughters, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No